CLINICAL TRIAL: NCT05883501
Title: Effect of Self-affirmation Versus Back Massage on Psychological Distress and Fear of Birth Among Primigravid Women in Third Trimester
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2252023
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Self-affirmation, Back Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Pregnant women will be given love cards containing positive affirmations that will be trained outside the classroom by asking the mother to practice alone once a day between waking up, before bed, or when relaxing.
  The suggestions will be implanted using simple language, easy to understand, in detail, and straightforward. For example, "From now, I know how to take care of myself in pregnancy and trust in my ability to birth my baby."
  Love cards will be developed through literature studies and expert tests containing positive affirmations for pregnancy and childbirth.
  Interventions: Behavioral: Self-affirmation versus back massage
- Group 2 (Experimental): The researcher will be used the heel of the hands, moving along the spine; using the palms moving hands with rocking movements from the top of the shoulder blade to the backbone; pressing fingertips, along both sides of the spine from the neck to the backbone and then stroking upward from the hip to the neck; stroking the shoulder muscles(trapezius); inching up the back, using fingertips placed on sides of spine, starting from the hipbone to the neck and then reversing the direction downward using fingertips in a raking fashion; massaging the lower back from the backbone across the waistline using the heel of the palm to make large circles; long gliding strokes from the hip up and over the shoulder (Nair ,. 2020 ; El-Hosary et al,. 2019).
  Back massage will be done in four sessions each session takes 10 minutes and will be performed every week.
  Interventions: Behavioral: Self-affirmation versus back massage

INTERVENTIONS:
Behavioral: Self-affirmation versus back massage — Self-affirmation is non-pharmacological intervention which represents structured sentences to convey to the subconscious mind to help in reprogramming negative thoughts into positive ones.
  Massage is defined as systematic touch of soft tissues for therapeutic purposes, such as pain relief, increased comfort and patient's relaxation

SUMMARY:
Based on the literature review, care must be emphasized on aspects of self-strengthening or self-affirmation to reduce stress and fear and equip women with the ability to manage stress and fear due to negative thoughts. Accordingly, the present study aimed to investigate and compare the effects of self-affirmation versus back massage on psychological distress and fear of birth among primigravid women in third trimester.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant women aged 20-35 years.

  * Primigravida women.
  * Read &write.
  * During third trimester of pregnancy.
  * Free from any medical, obstetric, gynecological and other psychological risk factors and /or conditions
  * With normal course of pregnancy.
  * Attend regular antenatal care visits.
  * With intact back skin and free from burn, wound or any scar, injury, inflammation and allergy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female pregnant women
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | 2 months
  The Kessler Psychological Distress Scale (K10) is a simple measure of psychological distress (Kessler et al., 2003). The K10 scale involves 10 questions about emotional states each with a five-level response scale. The measure can be used as a brief screen to identify levels of distress
Fear of childbirth | 2 months
  The Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) is a standardized screening method for measuring fear of childbirth during pregnancy (Wijma et al., 1998).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No